CLINICAL TRIAL: NCT03034278
Title: Improving Opioid Prescription Safety After Surgery
Brief Title: Self-reported Usage Patterns of Opioid Analgesic Medications After Surgery
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-1938; 1K23DA040923-01A1 (NIH)
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Opioid Use
Keywords: opioid use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post surgery patients: Patients prescribed with opioid analgesic medications following surgery.
  Interventions: Other: Not applicable - no intervention

INTERVENTIONS:
Other: Not applicable - no intervention — Not applicable - no intervention, observational survey study.

SUMMARY:
The primary objective of this study is to better understand post-discharge utilization of prescribed opioid analgesic medications following surgery. A secondary objective of this study is to gain a better understanding of prevailing modes of storage for opioid medications.

DETAILED DESCRIPTION:
Hypothesis:

Prescription of medications for analgesia after surgery frequently occurs on an empiric rather than individualized basis. The investigator will hypothesize that prescribed opioid medications for analgesia after discharge from the hospital / surgery center are frequently not taken.

Aims:

i) The descriptive first aim of this study is to define self-reported usage patterns of opioid analgesic medications at home following surgery.

ii) The descriptive second aim of this study is to define prevailing modes of storage and/or disposal for opioid medications prescribed to patients after hospital discharge following surgery.

iii) The analytical second aim of this study is to characterize patients who do not take significant amounts of their prescribed opioid medications.

Background & Exploratory Objective (s):

Accidents (unintentional injuries) were the 5th leading cause of death among the general population in the United States in 2010. Among persons 1-44 years of age accidents represented the leading cause of death. And, within this group, pharmaceuticals were the #1 course of death. Of the 22,134 medication associated deaths in 2010, 75.2% included opioid analgesics. The trajectory of this development is alarming: Deaths from prescription opioid overdoses have more than tripled in recent years. Of special concern is that children are especially vulnerable to unintentional medication overdosing, accounting for 71,224 annual emergency room visits for this reason from 2004-2005 alone. In addition to the individual burden from morbidity and mortality, the costs of prescription opioid abuse to society are immense: The average health care costs for patients abusing opioids are 8 times higher than for non-abusers. In the United States alone, $55.7 billion were spent on sequelae in the workplace and in healthcare costs. Accordingly, prescription drug overdosing has been coined "An American Epidemic" and increasing resources to tackle this rapidly growing public health problem have been made available on a national (National Institutes of Health, U.S. Food and Drug Administration) and the state level as part of the Colorado Consortium for Prescription Drug Abuse created through Governor Hickenlooper's efforts with the National Governors Association.

Additionally, the prescription of opioids following surgery usually occurs using a "one size fits all approach", leading potentially to many unused opioids that are then likely to be utilized in a fashion unintended by prescribing clinician.

The goal of the proposed study is to assess self-reported intake relative to prescribed amounts of analgesic medications after surgery. Better knowledge of this relationship will permit the design of tools to individualize analgesic pharmacotherapy after hospital discharge. The goal is to reduce the amount of opioid prescriptions that are not needed and to improve non-opioid analgesia.

These data will inform future studies to design more patient-centered opioid prescribing tools, which are based on anticipated need. This will likely decrease the amounts of prescribed opioids that are available for non-medical use. Future studies will be aimed to standardize their use to provide improved analgesia upon discharge following surgery.

ELIGIBILITY:
Inclusion Criteria:

Adult patients undergoing:

* Cesarean section,
* Gastrointestinal surgery, or
* Thoracic surgery.

Exclusion Criteria:

* Patients under the age of 18 years of age,
* Patients known or suspected to be pregnant at the time of discharge,
* Patients that are prisoners,
* Patients that are decisionally challenged,
* Patients that are blind, and
* Patients that are illiterate.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Design/Methods:
  Survey population: Patients ages 18-89 undergoing surgery at the University of Colorado Hospital are eligible. We will focus on patients after Cesarean section surgery, gastrointestinal, and thoracic surgery.
  Following exclusion of all patients under the age of 18 years, patients who do not understand Spanish or English, and patients returning to institutional settings (e.g. prison, jail, mental health facility), pregnant women, and decisionally challenged patients, the investigators will include all remaining patients in the sample.
  The investigators will focus on adult patients after 1) Cesarean section, 2) thoracic surgery procedures, and 3) gastrointestinal surgery procedures.
Sampling Method: Non-Probability Sample
Enrollment: 785 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Ratio of patient-reported intake of oral opioids to prescribed amount of oral opioid medications | 4 weeks after hospital discharge date.
  A self-report survey will assess opioid medication use in surgical patients during the 4 weeks following hospital discharge.

SECONDARY OUTCOMES:
Storage of opioid medication in surgical patients after hospital discharge | 4 weeks after hospital discharge date.
  A self-report survey will assess storage of opioid medication in surgical patients up to 4 weeks after discharge from the hospital.

OTHER OUTCOMES:
Description of surgical patients from their electronic medical record | Date of admission to hospital up to thirty days after hospital discharge date.
  For each surgical patient who completes the study survey we will access their electronic medical record and characterize them by age, gender, race, type of insurance, body mass index, comorbid medical conditions, type of surgical procedure and severity, pre-operative and in-hospital opioid use, and use of acetaminophen and NSAIDs. We will then relate these patient characteristics to the participants responses on the study surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Bartels, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Bartels K, Binswanger IA, Hopfer CJ. Sources of Prescription Opioids for Nonmedical Use. J Addict Med. 2016 Mar-Apr;10(2):134. doi: 10.1097/ADM.0000000000000192. No abstract available. PMID 26985647
- [Result] Carrico JA, Mahoney K, Raymond KM, McWilliams SK, Mayes LM, Mikulich-Gilbertson SK, Bartels K. Predicting Opioid Use Following Discharge After Cesarean Delivery. Ann Fam Med. 2020 Mar;18(2):118-126. doi: 10.1370/afm.2493. PMID 32152015
- [Result] Abrams BA, Murray KA, Mahoney K, Raymond KM, McWilliams SK, Nichols S, Mahmoudi E, Mayes LM, Fernandez-Bustamante A, Mitchell JD, Meguid RA, Zanotti G, Bartels K. Postdischarge Pain Management After Thoracic Surgery: A Patient-Centered Approach. Ann Thorac Surg. 2020 Nov;110(5):1714-1721. doi: 10.1016/j.athoracsur.2020.04.048. Epub 2020 Jun 1. PMID 32497643
- [Result] Bartels K, Mahoney K, Raymond KM, McWilliams SK, Fernandez-Bustamante A, Schulick R, Hopfer CJ, Mikulich-Gilbertson SK. Opioid and non-opioid utilization at home following gastrointestinal procedures: a prospective cohort study. Surg Endosc. 2020 Jan;34(1):304-311. doi: 10.1007/s00464-019-06767-1. Epub 2019 Apr 3. PMID 30945059

DOCUMENTS (1):
  • Informed Consent Form (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT03034278/ICF_000.pdf